CLINICAL TRIAL: NCT05943028
Title: Chief Physician of the Department of Anesthesiology of the Southern Theater General Hospital
Brief Title: Effect of Subanesthetic Dose Esketamine on Propofol-refentanil Closed-loop Targeted Controlled Infusion
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: bo xu (Other)
Responsible Party: Sponsor-Investigator, bo xu, professor, Guangzhou General Hospital of Guangzhou Military Command
Organization: Guangzhou General Hospital of Guangzhou Military Command (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Effects of esketamine on EEG
Record Dates: First submitted 2023-06-27; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Esketamine
Keywords: closed-loop TCI; Esketamine; general anesthesia; NI

STUDY DESIGN:
Intervention Model Description: The control group chose the original preset value of 36 as the baseline value of EEG closed-loop feedback guidance (derived from the team's previous research results.The experimental group selected the preset value of 36+N as the baseline value of the new EEG closed-loop feedback guidance (the N value was 6-8 from the pre-experiment).Samples that met the inclusion criteria were randomized and randomly included in the experimental and control groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants were assigned to the management and control groups, and neither group of researchers nor subjects was clear about their group. Data statistical analysts and clinical trial participants maintain independence in their work.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Experimental): The preset EEG value of 36 in closed-loop target-controlled infusion is the baseline value of EEG closed-loop feedback guidance (obtained by the team's previous research results)
  Interventions: Drug: Subanesthetic dose of esketamine
- Experimental group (Experimental): Due to the action of esketamine in closed-loop target-controlled infusion, the EEG preset value of 36+N is the baseline value of the new EEG closed-loop feedback guidance (pre-experiment and literature data, N value is 6-8)
  Interventions: Drug: Subanesthetic dose of esketamine

INTERVENTIONS:
Drug: Subanesthetic dose of esketamine — Both groups were given NI-guided propofol-refentanil dual-channel closed-loop target-controlled infusion under general anesthesia with a laryngeal mask/endotracheal intubation. The experimental group (EEG feedback index 36+N) and the control group (EEG feedback index 36) were intravenously injected esketamine 0.2mg∙kg-1 before anesthesia induction, followed by continuous 5μg∙kg-1∙min-1 infusion to maintain anesthesia for 30 minutes, and the maximum cumulative dose allowed was 100mg. In both groups, the infusion was stopped 30 minutes before the end of surgery.
  Other Names: Esketamine hydrochloride injection

SUMMARY:
The propofol-refentanil program-controlled closed-loop target-controlled infusion system based on NI guidance has been clinically verified. In the case of clinical use of esketamine, the separation anesthesia properties do not affect the accuracy and safety of closed-loop system guidance. However, whether the specific degree of impact can be quantified, and based on quantitative indicators, this model can be better applied to a wider range of clinical actual conditions and different drug administration backgrounds.

DETAILED DESCRIPTION:
The first phase is data collection on the effect of subanesthetic doses of esketamine on NI EEG in closed-loop target-controlled infusion systems for general anesthesia. According to the observation of pre-experiments and the latest literature at home and abroad, foreign studies have confirmed that esketamine does not affect the overall stability of the closed-loop system, and we verified the reliability of this conclusion through pre-experiments. In order to clarify the degree of influence of subanesthetic dose of esketamine on EEG, it is necessary to include a certain amount of esketamine applied to the anesthesia sample of closed-loop target controlled infusion system, through the main observation indicators: the change of EEG NI value after the administration of subanesthetic dose of esketamine during the anesthesia maintenance period, the change of EEG power spectrum, and the quantitative ratio change trend of brain waves (α, β, θ, δ waves). The difference in EEG NI value, power spectrum and dynamic transformation of brain wave increased due to the action of subanesthetic dose of esketamine was obtained, and the difference was quantified by the attribution of data to the degree of change of the actual EEG NI value. According to the preset guidance EEG NI value of the original closed-loop target-controlled infusion drug delivery system 36, the guidance preset value of the closed-loop system of 36+N in the clinical administration scenario of subanesthetic dose of esketamine was reset as the new EEG closed-loop feedback baseline.

The second phase is the validation of the effect of esketamine equivalent to the subanesthetic dose on closed-loop target-controlled infusion general anesthesia based on regulated NI(36+N) feedback.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients undergoing laparoscopic general anesthesia surgery with anesthesia duration > 60min, 2.18~55 years old, 3.BMI≥18.5kg/m2, 4. ASA Class I~II

Exclusion Criteria:

* Exclude patients with any of the following criteria:

  1. Contraindications to esketamine, propofol or refentanil;
  2. Allergic reactions to egg/soy products; Hypersensitivity to fentanyl analogues;
  3. Known/suspected neurological diseases, tumors, strokes, neurodegenerative diseases, severe head injuries, seizures, previous EEG abnormalities, cognitive deficits, acquired scalp/skull abnormalities, psychiatric diseases, severe depression, post-traumatic stress disorder, psychosis;
  4. Taking psychotropic drugs within the past 7 days,
  5. History of substance abuse/abuse or pregnancy in the past 30 days;
  6. Currently involved in any other research involving drugs or devices.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
EEG value | From the beginning to the end of the surgery, an average of 4 hours
  Differences in EEG values between the two groups based on different feedback baselines
Anesthesia maintains drug consumption | From the beginning to the end of the surgery, an average of 4 hours
  Two groups of propofol and refentanil consumption

SECONDARY OUTCOMES:
heart rate | From the beginning to the end of the surgery, an average of 4 hours
  Rate variations and differences throughout the process
Blood pressure | From the beginning to the end of the surgery, an average of 4 hours
  Changes and differences in blood pressure throughout the process
pulse | From the beginning to the end of the surgery, an average of 4 hours
  Changes and differences in pulse throughout the process

CONTACTS AND LOCATIONS:
Overall Officials: Shengchao Li, Graduate, Principal Investigator — The First Clinical College of Southern Medical University

IPD SHARING:
Plan to Share IPD: No
Data collection is recorded from anesthesia records in the original medical record and uploaded to Data Digital for sharing and management(https://www.bcg.com/publications/2022/how-to-build-a-data-and-digital-strategy)

REFERENCES:
- [Background] Liu N, Chazot T, Hamada S, Landais A, Boichut N, Dussaussoy C, Trillat B, Beydon L, Samain E, Sessler DI, Fischler M. Closed-loop coadministration of propofol and remifentanil guided by bispectral index: a randomized multicenter study. Anesth Analg. 2011 Mar;112(3):546-57. doi: 10.1213/ANE.0b013e318205680b. Epub 2011 Jan 13. PMID 21233500
- [Background] Napoleone G, van Heusden K, Cooke E, West N, Gorges M, Dumont GA, Ansermino JM, Merchant RN. The Effect of Low-Dose Intraoperative Ketamine on Closed-Loop-Controlled General Anesthesia: A Randomized Controlled Equivalence Trial. Anesth Analg. 2021 Nov 1;133(5):1215-1224. doi: 10.1213/ANE.0000000000005372. PMID 33560659